CLINICAL TRIAL: NCT05925686
Title: Tramadol Administered Orally to Healthy Subjects for the Improvement of Its Detection in Biological Matrices in the Context of Anti-Doping Control
Brief Title: Tramadol to Improve Its Detection in Biological Matrices in Anti-doping Controls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IMIMFCTL/TRAM/1
Record Dates: First submitted 2023-05-15; First posted 2023-06-29 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-03

CONDITIONS: Healthy
MeSH Terms: interventions — Tramadol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tramadol. (Experimental)
  Interventions: Drug: Tramadol.

INTERVENTIONS:
Drug: Tramadol. — Orally single dose administration of Tramadol 75 mg for ultra-rapid metabolizers and 100 mg for extensive and poor metabolizers.

SUMMARY:
Orally single dose administration of Tramadol 75 mg for ultra-rapid metabolizers and 100 mg for extensive and poor metabolizers will be administered with the objective to evaluate urine and blood concentrations in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 55 years.
* Weight ≥ 50 kg and ≤ 100 kg.
* Body mass index (BMI) ≥ 18 and ≤ 30.
* Negative serum pregnancy test (women only).
* Signed informed consent prior to any study-mandated procedure.

Exclusion Criteria:

* Smoker of more than 5 cigarettes per day in the last 3 months prior to participate in the study.
* History of psychiatric disorders, alcoholism or drug abuse.
* Positive urine pregnancy test.
* No highly effective anticonception measures during the trial.
* Breastfeeding.
* Positive blood or urine test for drugs of abuse or alcohol breath test prior to study drug administration.
* Any clinically relevant disease or condition (cardiovascular, renal, hepatic, endocrine, hematology, neurology o other acute or chronic diseases) that in the judgment of the investigator might interfere with the subject's ability to comply with study procedures or requirements and/or bias the interpretation of the study results and/or jeopardize the subject's safety.
* Major Surgery last 6 months.
* Ongoing gastrointestinal diseases or history of gastrointestinal surgery affecting absorption.
* Subjects with a clinically significant disease within one month prior to study drug administration.
* Any clinically relevant findings in physical examination, vital signs, 12-lead ECG and safety laboratory parameters.
* Positive hepatitis or HIV test.
* Known hypersensitivity to any drug or drug excipients.
* Use of drugs known to induce or inhibit hepatic drug metabolism within one month prior to study administration or during the study and use of citrus juice during the study.
* Any prescription or over-the-counter (OTC) product including herbal, homeopathic, vitamins, minerals and nutritional supplements within 2 weeks prior to study drug administration.
* Intake of more than 5 units per day of beverages containing xanthine (coffee, tea or cola drinks).
* Donation of blood or plasma within one month prior to study drug administration or transfusion of blood or plasma for medical/surgical reasons or intention to donate blood or plasma within one month after study drug administration.
* History of inadequate venous access and/or experience of difficulty donating blood.
* Not able/not willing to accept restrictions regarding diet, physical exercise, and consumption of alcohol and/or xanthine containing items when out of CRU.
* Subject included in a clinical study within 3 months prior to study drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Urine concentration on Tramadol. | From baseline to 8 hours.

SECONDARY OUTCOMES:
Plasma and dried blood spots (DBS) concentration on Tramadol. | From baseline to 12 hours.

OTHER OUTCOMES:
Adverse effects. | From baseline to 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- IMIM (Institut Hospital del Mar d'Investigacions Mèdiques), Barcelona, Spain